CLINICAL TRIAL: NCT02624180
Title: Inflammatory Pathogenesis of Coronary Atherosclerosis in HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00070892; 1R01HL125059 (NIH)
Record Dates: First submitted 2015-11-11; First posted 2015-12-08 (Estimated); Results first posted 2021-08-19 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease; Human Immunodeficiency Virus
MeSH Terms: conditions — Coronary Artery Disease; Acquired Immunodeficiency Syndrome | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colchicine (Experimental): Colchicine 0.6 mg daily by mouth
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Placebo for colchicine 1 tablet by mouth daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Administered to determine the effect of anti-inflammatory agents on coronary and systemic endothelial function in patients with coronary artery disease.
  Other Names: Colcrys
  Arms: Colchicine
Drug: Placebo — A substance containing no medication
  Arms: Placebo

SUMMARY:
The investigators are studying whether an anti-inflammatory intervention improves impaired coronary endothelial function (CEF) in HIV+ people with no clinical coronary artery disease (CAD).

DETAILED DESCRIPTION:
Survival in people with HIV has significantly improved with the use of antiretroviral therapy (ART) but HIV+ people now experience an increasing burden of chronic diseases, including coronary atherosclerosis and coronary artery disease (CAD). HIV patients manifest an increased risk of CAD and its consequences possibly due to interplay of inflammation with traditional risk factors (smoking, high cholesterol, and poor diet), some of the latter accentuated by ART.

What the investigators are studying in this program is the function of the coronary arteries and in particular the inner lining of the arteries called the endothelium in patients with HIV. The endothelium has several important functions; one of them is that under conditions of stress it releases a substance called nitric oxide which increases the size of the artery and increases blood flow. When it is not functioning normally the artery does not increase as much and blood flow does not increase during stress.

The investigators study coronary artery function with magnetic resonance imaging, or MRI. MRI is a method of obtaining images of what is happening inside the body. MRI does not involve radiation, x-ray, or injection of contrast. The investigators can measure flow in the artery and the dimension of the artery at rest and with a handgrip stress and learn the extent to which the artery dilates and flow increases with the stress. The investigators believe that inflammation can interfere with normal function and that by decreasing inflammation abnormal endothelial function may be improved.

Colchicine is an anti-inflammatory agent approved by the Food and Drug Administration (FDA) to treat arthritis and some other conditions. This drug is not approved for use to suppress inflammation in patients with coronary artery disease and improve coronary artery endothelial function. The FDA is allowing the use of colchicine or a placebo in this research study.

This study will involve 24 weeks of colchicine or placebo and 3 Magnetic Resonance Imaging (MRI) scans of the heart and other study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender who are 21 years of age (no upper age limit), HIV positive and taking stable ART (no change in ART regimen in last 3 months),
* HIV viral load <100 copies/mL (plasma HIV RNA concentration),
* Abnormal CEF at baseline (<7ml/min change in CBF during IHE as compared to resting value).

Exclusion Criteria:

* Patients unable to understand the risks, benefits, and alternatives of participation and give meaningful consent,
* Patients with contraindications to MRI such as implanted metallic objects (pre-existing cardiac pacemakers, cerebral clips) or indwelling metallic projectiles,
* History of clinical CAD, including acute coronary syndrome, myocardial infarction or revascularization,
* Resting ECG with evidence of Q wave myocardial infarction,
* Pregnant women,
* Recent history, within the past 3 months, of cocaine or heroin use,
* Moderate or greater renal impairment (estimated glomerular filtration rate <45ml/min),
* Moderate-severe hepatic disease (elevation in hepatic transaminases >3x upper limit of normal),
* Leukopenia (<3000/mm3) or thrombocytopenia (<100,000/mm3),
* CD4<200 cell/mm3,
* Chronic inflammatory condition such as lupus or rheumatoid arthritis, ulcerative colitis or Crohn's disease,
* Requirement for, or intolerance to, colchicine,
* Women of childbearing potential (even if using oral contraceptive agents) or intention to breastfeed,
* Chronic, continuous use of oral or IV steroid therapy or other immunosuppressive or biologic response modifiers or anti-inflammatory agents (chronic NSAIDs or acetylsalicylic acid (ASA) >81mg daily),
* History of chronic pericardial effusion, pleural effusion, ascites or peripheral neuropathy manifested by both signs and symptoms,
* Taking protease inhibitors (PI), cobicistat, or CYP3A4 inhibitors.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-11; Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Weiss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deanfield JE, Halcox JP, Rabelink TJ. Endothelial function and dysfunction: testing and clinical relevance. Circulation. 2007 Mar 13;115(10):1285-95. doi: 10.1161/CIRCULATIONAHA.106.652859. No abstract available. PMID 17353456
- [Background] Widlansky ME, Gokce N, Keaney JF Jr, Vita JA. The clinical implications of endothelial dysfunction. J Am Coll Cardiol. 2003 Oct 1;42(7):1149-60. doi: 10.1016/s0735-1097(03)00994-x. PMID 14522472
- [Background] Hays AG, Hirsch GA, Kelle S, Gerstenblith G, Weiss RG, Stuber M. Noninvasive visualization of coronary artery endothelial function in healthy subjects and in patients with coronary artery disease. J Am Coll Cardiol. 2010 Nov 9;56(20):1657-65. doi: 10.1016/j.jacc.2010.06.036. PMID 21050976
- [Background] Hays AG, Stuber M, Hirsch GA, Yu J, Schar M, Weiss RG, Gerstenblith G, Kelle S. Non-invasive detection of coronary endothelial response to sequential handgrip exercise in coronary artery disease patients and healthy adults. PLoS One. 2013;8(3):e58047. doi: 10.1371/journal.pone.0058047. Epub 2013 Mar 11. PMID 23536782
- [Background] Hays AG, Kelle S, Hirsch GA, Soleimanifard S, Yu J, Agarwal HK, Gerstenblith G, Schar M, Stuber M, Weiss RG. Regional coronary endothelial function is closely related to local early coronary atherosclerosis in patients with mild coronary artery disease: pilot study. Circ Cardiovasc Imaging. 2012 May 1;5(3):341-8. doi: 10.1161/CIRCIMAGING.111.969691. Epub 2012 Apr 5. PMID 22492483
- [Background] Nidorf SM, Eikelboom JW, Budgeon CA, Thompson PL. Low-dose colchicine for secondary prevention of cardiovascular disease. J Am Coll Cardiol. 2013 Jan 29;61(4):404-410. doi: 10.1016/j.jacc.2012.10.027. Epub 2012 Dec 19. PMID 23265346
- [Background] Brown BG, Lee AB, Bolson EL, Dodge HT. Reflex constriction of significant coronary stenosis as a mechanism contributing to ischemic left ventricular dysfunction during isometric exercise. Circulation. 1984 Jul;70(1):18-24. doi: 10.1161/01.cir.70.1.18. PMID 6426817
- [Derived] Bagchi S, Kwapong YA, Schar M, Bonanno G, Streeb V, Lai S, Gerstenblith G, Weiss RG, Hays AG. The Relationship Between Impaired Coronary Endothelial Function and Systemic Markers of Inflammation in People Living With HIV. J Acquir Immune Defic Syndr. 2023 May 1;93(1):47-54. doi: 10.1097/QAI.0000000000003162. PMID 36634369
- [Derived] Hays AG, Schar M, Barditch-Crovo P, Bagchi S, Bonanno G, Meyer J, Afework Y, Streeb V, Stradley S, Kelly S, Anders NM, Margolick JB, Lai S, Gerstenblith G, Weiss RG. A randomized, placebo-controlled, double-blinded clinical trial of colchicine to improve vascular health in people living with HIV. AIDS. 2021 Jun 1;35(7):1041-1050. doi: 10.1097/QAD.0000000000002845. PMID 33587443

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants randomized to colchicine withdrew before receiving study drug.
Period: Overall Study
Arm/Group | Colchicine | Placebo
Started | 43 | 38
Completed (Participants completing primary endpoint at 8 weeks) | 37 | 34
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colchicine | Placebo | Total
Number analyzed (Participants) | 43 | 38 | 81
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 54.66 [45.0 to 60.7] | 52.0 [45.2 to 57.4] | 54.25 [45.1 to 59.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 34 | 30 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 41 | 37 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 26 | 59
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Coronary Endothelial Function Measured by Percent Change in Coronary Blood Flow With Exercise (%) at 8 Weeks
Description: Percent change in coronary blood flow (CBF) from rest to that during isometric handgrip exercise (IHE) stress at 8 weeks.
Time Frame: Difference between measurements at baseline compared to measurement at 8 weeks
Measure: Mean (Standard Deviation); unit: Percent change from rest measurement
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 37 | 34
Percent change from rest measurement | 8.1 (4.4) | 13.4 (4.0)

2. Secondary Outcome: Coronary Endothelial Function at 24 Weeks;
Description: Change in coronary blood flow (CBF) from rest to that during isometric handgrip exercise (IHE) stress at 24 weeks.
Time Frame: At 24 weeks.
Measure: Median (Inter-Quartile Range); unit: Percent change from rest measurement
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 34 | 32
Percent change from rest measurement | -1.27 [-11.56 to 20.35] | 16.60 [-2.04 to 29.66]

3. Secondary Outcome: Change in Coronary Artery Cross-sectional Area (CSA) at 8 Weeks
Description: Change in CSA as measured by the difference between CSA at rest and under IHE stress at 8 weeks
Time Frame: Difference between measurements at baseline compared to measurement at 8 weeks
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline measurement
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 37 | 34
Percent change from baseline measurement | -0.10 [-5.75 to 3.99] | 1.53 [-3.76 to 6.63]

4. Secondary Outcome: Change in Coronary Artery Cross-sectional Area (CSA) at 24 Weeks
Description: Change in CSA as measured by the difference between CSA at rest and under IHE stress at 24 weeks
Time Frame: At 24 weeks
Measure: Median (Inter-Quartile Range); unit: Percent change from rest measurement
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 34 | 33
Percent change from rest measurement | -0.96 [-5.86 to 6.61] | 5.04 [-1.60 to 13.37]

5. Secondary Outcome: High-sensitivity C-reactive Protein (hsCRP) at 8 Weeks.
Description: High-sensitivity C-reactive protein (hsCRP) at 8 weeks
Time Frame: At 8 weeks.
Measure: Median (Inter-Quartile Range); unit: mg/l
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 37 | 34
mg/l | 1.65 [0.77 to 4.67] | 1.26 [0.86 to 2.68]

6. Secondary Outcome: Brachial Flow Mediated Dilatation (FMD) at 8 Weeks.
Description: Brachial flow mediated dilatation (FMD) at 8 weeks.
Time Frame: At 8 weeks
Measure: Median (Inter-Quartile Range); unit: % brachial artery dilation
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 37 | 34
% brachial artery dilation | 4.26 [1.76 to 6.17] | 4.12 [2.09 to 6.16]

7. Secondary Outcome: Interleukin-6 (IL-6) at 8 Weeks
Description: Interleukin-6 (IL-6) at 8 weeks
Time Frame: At 8 weeks
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 37 | 34
pg/ml | 0.53 [0.43 to 0.81] | 0.64 [0.42 to 0.85]

8. Secondary Outcome: High-sensitivity C-reactive Protein (hsCRP) at 24 Weeks
Description: High-sensitivity C-reactive Protein (hsCRP) at 24 weeks
Time Frame: At 24 weeks
Measure: Median (Inter-Quartile Range); unit: mg/l
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 35 | 32
mg/l | 1.00 [0.50 to 3.20] | 1.30 [0.80 to 2.20]

9. Secondary Outcome: Brachial Flow Mediated Dilatation (FMD) at 24 Weeks.
Description: Brachial Flow Mediated Dilatation (FMD) at 24 Weeks.
Time Frame: At 24 weeks
Measure: Median (Inter-Quartile Range); unit: % brachial artery dilation
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 30 | 30
% brachial artery dilation | 3.82 [2.25 to 7.25] | 3.46 [1.41 to 8.29]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over study enrollment (up to 24 weeks after randomization to study drug)
Description: Two participants randomized to colchicine withdrew before receiving study drug so number of participants at risk listed here as 41.
Arm/Group | Colchicine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/41 | 2/38
Other Adverse Events (participants affected / at risk) | 39/41 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine (N=41) | Placebo (N=38)
Hospitalization (Renal and urinary disorders) | 0 (0) | 1 (1) — Urinary tract infection requiring hospitalization
Hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1) — Participant underwent elective carotid endarterectomy during study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine (N=41) | Placebo (N=38)
Infection (Infections and infestations) | 9 (9) | 19 (19)
Gastrointestinal disorder (Gastrointestinal disorders) | 12 (12) | 9 (9)
Joint/Muscle Soreness/Stiffness (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9)
Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Extremity swelling (General disorders) | 0 (0) | 1 (1)
Dental pain/infection (General disorders) | 0 (0) | 3 (3)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Vision (Eye disorders) | 1 (1) | 0 (0)
Physical Injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Increased Aspartate Amino Trans (Hepatobiliary disorders) | 7 (7) | 6 (6)
Increased Alanine Amino Trans (Hepatobiliary disorders) | 7 (7) | 5 (5)
Decreased White Blood Cell (Blood and lymphatic system disorders) | 7 (7) | 4 (4)
Decreased Hematocrit (Blood and lymphatic system disorders) | 10 (10) | 8 (8)
Decreased Estimated GFR (Renal and urinary disorders) | 10 (10) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT02624180/Prot_SAP_000.pdf